CLINICAL TRIAL: NCT02209506
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Sequential-Cohort, Ascending Multiple Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MLN3126 in Healthy Non-Japanese and Japanese Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MLN3126 in Healthy Japanese and Non-Japanese Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Long-term animal toxicology findings (see detailed description).
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN3126_103; U1111-1156-8528 (Other: World Health Organziation)
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
Keywords: MLN3126

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Cohort 1A: MLN3126 100 mg Non-Japanese Participants (Experimental): MLN3126 100 mg, administered orally as tablets once on Day 1, followed by a 7 day washout period, followed by once daily administration for 7 days (Days 9 through 15) in healthy, non-Japanese participants.
  Interventions: Drug: MLN3126
- Cohort 2A: MLN3126 300 mg Non-Japanese Participants (Experimental): MLN3126 300 mg, administered orally as tablets, orally, once on Day 1, followed by a 7 day washout period, followed by once daily administration for 7 days (Days 9 through 15) in healthy, non-Japanese participants.
  Interventions: Drug: MLN3126
- Cohort 3A: MLN3126 800 mg Non-Japanese Participants (Experimental): MLN3126 800 mg, administered orally as tablets once on Day 1, followed by a 7 day washout period, followed by once daily administration for 7 days (Days 9 through 15) in healthy, non-Japanese participants.
  Interventions: Drug: MLN3126
- Cohort 4A: MLN3126 TBD Non-Japanese Participants (Experimental): The MLN3126 dose for this Cohort will be determined based on data collected from Cohort 3A. MLN3126, tablets, administered orally, once on Day 1, followed by a 7 day washout period, followed by once daily administration for 7 days (Days 9 through 15) in healthy, non-Japanese participants.
  Interventions: Drug: MLN3126
- Cohorts 1A - 4A: Matched Placebo Non-Japanese Participants (Experimental): MLN3126 placebo-matching tablets, administered orally, once on Day 1, followed by a 7 day washout period, followed by once daily administration for 7 days (Days 9 through 15) in healthy, non-Japanese participants.
  Interventions: Drug: MLN3126 Matched Placebo
- Cohort 1B: MLN3126 100 mg Japanese Participants (Experimental): MLN3126 100 mg, administered orally as tablets, once on Day 1, followed by a 7 day washout period, followed by once daily administration for 7 days (Days 9 though 15) in healthy, Japanese participants.
  Interventions: Drug: MLN3126
- Cohort 2B: MLN3126 300 mg Japanese Participants (Experimental): MLN3126 300 mg, administered orally as tablets, once on Day 1, followed by a 7 day washout period, followed by once daily administration for 7 days (Days 9 through 15) in healthy, Japanese participants.
  Interventions: Drug: MLN3126
- Cohort 3B: MLN3126 800 mg Japanese Participants (Experimental): MLN3126 800 mg, tablets, orally, once on Day 1, followed by a 7 day washout period, followed by MLN3126 800 mg, tablets, orally, once daily for 7 days (Days 9 through 15) in healthy, Japanese participants.
  Interventions: Drug: MLN3126
- Cohort 4B: MLN3126 TBD Japanese Participants (Experimental): The MLN3126 dose for this Cohort will be determined based on data collected from Cohort 3B. MLN3126, tablets, administered orally, once on Day 1, followed by a 7 day washout period, followed by once daily administration for 7 days (Days 9 through 15) in healthy, Japanese participants.
  Interventions: Drug: MLN3126
- Cohorts 1B - 4B: Matched Placebo Japanese Participants (Experimental): MLN3126 placebo-matching tablets, administered orally, once on Day 1, followed by a 7 day washout period, followed by once daily for 7 days (Days 9 through 15) in healthy, Japanese participants.
  Interventions: Drug: MLN3126 Matched Placebo

INTERVENTIONS:
Drug: MLN3126 — MLN3126 tablets
  Arms: Cohort 1A: MLN3126 100 mg Non-Japanese Participants; Cohort 1B: MLN3126 100 mg Japanese Participants; Cohort 2A: MLN3126 300 mg Non-Japanese Participants; Cohort 2B: MLN3126 300 mg Japanese Participants; Cohort 3A: MLN3126 800 mg Non-Japanese Participants; Cohort 3B: MLN3126 800 mg Japanese Participants; Cohort 4A: MLN3126 TBD Non-Japanese Participants; Cohort 4B: MLN3126 TBD Japanese Participants
Drug: MLN3126 Matched Placebo — MLN3126 placebo-matching tablets
  Arms: Cohorts 1A - 4A: Matched Placebo Non-Japanese Participants; Cohorts 1B - 4B: Matched Placebo Japanese Participants

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single and multiple oral dosing of MLN3126 in ascending doses in healthy non-Japanese and Japanese participants.

DETAILED DESCRIPTION:
MLN3126 is being tested to find a safe and well-tolerated dose in healthy people and to assess how MLN3126 is processed by the body. In total, approximately 64 participants will be enrolled in the study.

This study is composed of 2 parts: Part A healthy non-Japanese participants and Part B healthy Japanese participants. Each part will consist of 4 Cohorts with 8 participants in each Cohort. In each Cohort, 6 participants will receive MLN3126 and 2 participants will receive matched placebo within 30 minutes after the start of a standard breakfast. The starting dose will be 100 mg followed by doses of 300 mg, 800 mg, and a dose to be determined during the study. Progression to the next dose level will only occur if the previous dose level was considered to be safe and well tolerated.

This single-center trial will be conducted in the United States. The overall time to participate in this study is up to 20 days. All participants will be contacted by telephone 7 days after the last dose of study drug for a follow-up assessment.

Due to toxicology findings from a long-term animal study, Takeda made the decision to terminate this study. No clinically significant safety and/or tolerability issues have been observed or reported in participants exposed to MLN3126.

ELIGIBILITY:
Inclusion Criteria:

Part A (Healthy non-Japanese participants):

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures, including requesting that a participant fast for any laboratory evaluations.
3. Is a male or female adult, 18 to 55 years of age, inclusive, at the time of informed consent and study drug dosing.
4. Is a healthy adult male or female participant as evidenced by their medical history, complete physical examination, vital signs, electrocardiogram (ECG), and safety laboratory evaluations.
5. Weighs at least 45 kg and has a body mass index (BMI) between 18 and 30 kg/m^2 inclusive at Screening.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of informed consent throughout the duration of the study to their next postconfinement menstruation. In addition, participants must be advised not to donate ova during this period.

Part B (Healthy Japanese participants):

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures, including requesting that a participant fast for any laboratory evaluations.
3. Is a male or female adult, 20 to 55 years of age, inclusive, at the time of informed consent and study drug dosing, is of Japanese descent (born to Japanese parents and grandparents and has lived outside Japan for less than 15 years), and maintains a Japanese diet and lifestyle.
4. Is a healthy adult male or female participant as evidenced by their medical history, complete physical examination, vital signs, ECG, and safety laboratory evaluations.
5. Weighs at least 45 kg and has a BMI between 18 and 28 kg/m^2 inclusive at Screening.
6. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after the last dose.
7. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to routinely use adequate contraception from signing of informed consent throughout the duration of the study to their next postconfinement menstruation. In addition, participants must be advised not to donate ova during this period.

Exclusion Criteria:

Part A (Healthy non-Japanese participants) and Part B (Healthy Japanese participants):

1. Has received any investigational compound within 30 days or 5 half-lives of the investigational compound, whichever is longer, prior to the first dose of study medication.
2. Has received MLN3126 in a previous clinical study.
3. Is an immediate family member, study site employee, or in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. Has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal (GI), or endocrine disease or allergic skin rash or other abnormality which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of MLN3126.
6. Has a positive urine drug result for drugs of abuse at Screening or Check-in (Day -1).
7. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse (defined as 4 or more alcoholic beverages per day) within 1 year prior to the Screening Visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
8. Has taken any excluded medication, supplements, or food products listed in the Excluded Medications and Dietary Products section of the protocol.
9. If female, the participant is pregnant or lactating or intending to become pregnant before or during the study, including the timeframe to the participant's next post-confinement menstruation after participating in this study.
10. If male, the participant intends to donate sperm during the course of this study or for 12 weeks thereafter.
11. Has current or recent (within 6 months) GI disease that would be expected to influence the absorption of drugs (ie, a history of malabsorption, any surgical intervention known to impact absorption [eg, bariatric surgery or bowel resection], esophageal reflux, peptic ulcer disease, erosive esophagitis, or frequent [more than once per week] occurrence of heartburn).
12. Has Gilbert's syndrome or bilirubin level 1.2x the upper limits of normal (ULN).
13. Has a history of cancer, except basal cell carcinoma, that has been in remission for at least 5 years prior to Day 1.
14. Has a positive test result for hepatitis B surface antigen (HBsAg) or antibody to hepatitis C virus (anti-HCV) at Screening or a known history of human immunodeficiency virus infection.
15. Has used nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patch or nicotine gum) within 28 days prior to Check-in (Day -1). Cotinine test is positive at Screening or Check-in (Day -1).
16. Has poor peripheral venous access.
17. Has donated or lost 450 mL or more of his or her blood volume (including plasmapheresis) or had a transfusion of any blood product within 45 days prior to Day 1.
18. Has a Screening or Check-in (Day -1) abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator.
19. Has a QT interval with Fridericia correction method (QTcF) > 430 milliseconds (ms) for men or > 450 ms for women or a PR outside the range of 120 to 210 ms confirmed upon repeat testing within a maximum of 30 minutes, at the Screening Visit or Check-in (Day -1).
20. Has abnormal Screening or Check-in (Day -1) laboratory values that suggest a clinically significant underlying disease or participant with the following laboratory abnormalities: Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 1.5 ULN.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Neptune City, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at single site in the United States from 04 August 2014 to 09 December 2014.
Pre-assignment Details: Part A was performed on non-Japanese participants and Part B was performed on Japanese participants. Planned doses of MLN3126 800 mg to be decided (TBD) dose for Part A, and MLN3126 300 mg, 800 mg, and TBD dose for Part 2 were not administered due to early termination of the study.
Groups:
- Part A: Placebo; Part B: Placebo: MLN3126 placebo-matching tablet, orally, once on Day 1 of the single dosing period, followed by 1 week washout period, further followed by MLN3126 placebo-matching tablets, orally, once daily from Day 9 up to Day 15 of the 7 day multiple dosing period.
- Part A: MLN3126 100 mg; Part B: MLN3126 100 mg: MLN3126 100 mg, tablet, orally, once on Day 1 of the single dosing period, followed by 1 week washout period, further followed by MLN3126 100 mg, tablets, orally, once daily from Day 9 up to Day 15 of the 7 day multiple dosing period.
- Part A: MLN3126 300 mg: MLN3126 300 mg, tablet, orally, once on Day 1 of the single dosing period, followed by 1 week washout period, further followed by MLN3126 300 mg, tablets, orally, once daily from Day 9 up to Day 15 of the 7 day multiple dosing period.
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: Placebo | Part B: MLN3126 100 mg
Started | 3 | 6 | 6 | 2 | 6
Completed | 3 | 6 | 6 | 2 | 5
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis set included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: Placebo | Part B: MLN3126 100 mg | Total
Number analyzed (Participants) | 3 | 6 | 6 | 2 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (7.77) | 38.8 (12.91) | 36.3 (7.12) | 52.5 (0.71) | 41.0 (12.47) | 39.7 (10.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 0 | 3 | 8
  Male | 1 | 4 | 5 | 2 | 3 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 1 | 1 | 4 | 0 | 0 | 6
  Non Hispanic or Latino | 2 | 5 | 2 | 2 | 6 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 2 | 6 | 9
  Black or African American | 2 | 3 | 2 | 0 | 0 | 7
  White | 1 | 2 | 3 | 0 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 6 | 2 | 6 | 23
Height [Mean (Standard Deviation); unit: centimeter] | 173.3 (4.93) | 173.0 (14.71) | 170.3 (10.84) | 170.0 (5.66) | 163.2 (9.33) | 169.5 (10.76)
Weight [Mean (Standard Deviation); unit: kilogram] | 81.70 (13.023) | 82.50 (15.920) | 79.50 (13.435) | 74.45 (3.323) | 64.15 (10.227) | 76.12 (14.004)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter] | 27.13 (3.616) | 27.36 (2.080) | 27.25 (2.547) | 25.77 (0.564) | 23.94 (1.559) | 26.27 (2.531)
Smoking Classification [Number; unit: participants]
  Never Smoked | 2 | 5 | 4 | 1 | 4 | 16
  Ex-Smoker | 1 | 1 | 2 | 1 | 2 | 7
Xanthine/Caffeine History [Number; unit: participants]
  Consumer | 0 | 2 | 0 | 1 | 4 | 7
  Non-Consumer | 3 | 4 | 6 | 1 | 2 | 16
Female Reproductive Status [Number; unit: participants] — This baseline characteristic was analyzed only in female participants.
  participants
    Postmenopausal | 0 | 0 | 0 | 0 | 1 | 1
    Surgically Sterile | 0 | 1 | 0 | 0 | 0 | 1
    Female of Childbearing Potential | 2 | 1 | 1 | 0 | 2 | 6
Alcohol Classification [Number; unit: participants]
  Never Drunk | 1 | 4 | 2 | 0 | 0 | 7
  Current Drinker | 2 | 1 | 3 | 2 | 6 | 14
  Ex-Drinker | 0 | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline up to 7 days after last dose of study drug (Day 22)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Part A: Placebo | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: Placebo | Part B: MLN3126 100 mg
Number analyzed (Participants) | 3 | 6 | 6 | 2 | 6
participants | 1 | 1 | 1 | 0 | 2

2. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Electrocardiogram Measurements at Least Once Post Dose
Description: A standard 12-lead ECG was performed. The percentage of participants with markedly abnormal electrocardiogram (ECG) findings during the study.
Time Frame: Baseline up to 7 days after last dose of study drug (Day 22)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Placebo | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: Placebo | Part B: MLN3126 100 mg
Number analyzed (Participants) | 3 | 6 | 6 | 2 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests at Least Once Post Dose
Description: The percentage of participants with any markedly abnormal, according to Takeda criteria, standard safety laboratory values, including hematology, serum chemistry, and urinalysis, during the treatment period.
Time Frame: Baseline up to 7 days after last dose of study drug (Day 22)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Placebo | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: Placebo | Part B: MLN3126 100 mg
Number analyzed (Participants) | 3 | 6 | 6 | 2 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Percentage of Participants Who Meet the Markedly Abnormal Criteria for Vital Sign Measurements at Least Once Post Dose
Description: The percentage of participants who meet markedly abnormal criteria designated by Takeda Global Research and Development Center, Inc. (TGRD). Criteria for markedly abnormal vital signs included body temperature, systolic blood pressure, diastolic blood pressure and pulse rate.
Time Frame: Baseline up to 7 days after last dose of study drug (Day 22)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Placebo | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: Placebo | Part B: MLN3126 100 mg
Number analyzed (Participants) | 3 | 6 | 6 | 2 | 6
percentage of participants | 3 | 2 | 6 | 0 | 8

5. Secondary Outcome: Cmax: Maximum Plasma Concentration for MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who received the study drug and had at least 1 measurable plasma concentration for either MLN3126 or its M-I metabolite.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
nanogram per milliliter (ng/mL)
  Day 1 (MLN3126) (n=6, 6, 6) | 2053.33 (420.983) | 3220.00 (730.479) | 2526.67 (702.244)
  Day 15 (MLN3126) (n=6, 6, 5) | 1845.00 (617.665) | 3088.33 (721.565) | 2200.00 (541.618)
  Day 1 (M-I) (n=6, 6, 6) | 167.00 (73.645) | 225.77 (74.661) | 157.60 (83.847)
  Day 15 (M-I) (n=6, 6, 5) | 149.57 (79.078) | 176.58 (55.561) | 149.12 (80.138)

6. Secondary Outcome: Tmax- Time to Reach the Cmax for MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: The PK analysis set included all participants who received the study drug and had at least 1 measurable plasma concentration for either MLN3126 or its M-I metabolite.
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Day 1 (MLN3126) (n=6, 6, 6) | 4.00 [2.0 to 4.0] | 4.00 [4.00 to 4.00] | 4.00 [4.00 to 4.00]
  Day 15 (MLN3126) (n=6, 6, 5) | 4.00 [2.0 to 4.0] | 4.00 [2.0 to 4.0] | 4.00 [4.00 to 4.00]
  Day 1 (M-I) (n=6, 6, 6) | 5.00 [4.0 to 8.0] | 6.00 [4.0 to 8.0] | 6.00 [4.0 to 6.0]
  Day 15 (M-I) (n=6, 6, 5) | 6.00 [4.0 to 6.0] | 4.00 [4.00 to 4.00] | 4.00 [4.0 to 8.0]

7. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau for MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL
  Day 1 (MLN3126) (n=6, 6, 6) | 21429.42 (3241.902) | 41451.93 (10339.782) | 27344.25 (6318.106)
  Day 15 (MLN3126) (n=6, 6, 5) | 15748.80 (3632.489) | 26353.06 (5626.212) | 18166.90 (4516.041)
  Day 1 (M-I) (n=6, 6, 6) | 2027.06 (1038.274) | 2935.78 (1180.471) | 1721.86 (768.842)
  Day 15 (M-I) (n=6, 6, 5) | 1698.10 (857.178) | 1920.06 (689.354) | 1634.08 (849.800)

8. Secondary Outcome: AUC (0-last): Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL
  Day 1 (MLN3126) (n=6, 6, 6) | 28827.86 (4652.165) | 55970.97 (14936.883) | 35900.38 (8806.878)
  Day 15 (MLN3126) (n=6, 6, 5) | 19240.50 (4032.308) | 33136.84 (7352.192) | 22929.63 (6521.723)
  Day 1 (M-I) (n=6, 6, 6) | 2467.13 (1308.583) | 3713.57 (1628.713) | 2025.77 (888.467)
  Day 15 (M-I) (n=6, 6, 5) | 2017.37 (989.383) | 2392.01 (930.338) | 1989.59 (1005.862)

9. Secondary Outcome: AUC(0-96): Area Under the Plasma Concentration-time Curve From Time 0 to 96 Hours Post Dose for MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL
  Day 1 (MLN3126) (n=6, 6, 6) | 28827.86 (4652.165) | 55971.02 (14936.843) | 35900.38 (8806.878)
  Day 15 (MLN3126) ((n=6, 6, 5) | 19240.50 (4032.308) | 33136.80 (7352.169) | 22929.63 (6521.723)
  Day 1 (M-I) (n=6, 6, 6) | 2478.39 (1296.387) | 3726.75 (1616.928) | 2051.37 (885.185)
  Day 15 (M-I) (n=6, 6, 5) | 2042.91 (995.133) | 2413.78 (935.159) | 2010.24 (993.327)

10. Secondary Outcome: AUC (0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: predose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
ng*hr/mL
  Day 1 (MLN3126) (n=6, 6, 6) | 29005.04 (4679.572) | 56338.09 (15089.327) | 36073.07 (8916.201)
  Day 15 (MLN3126) (n=6, 6, 5) | 19328.57 (4036.507) | 33250.14 (7370.421) | 23046.44 (6603.581)
  Day 1 (M-I) (n=6, 6, 6) | 2499.49 (1304.091) | 3747.82 (1631.659) | 2065.18 (892.563)
  Day 15 (M-I) (n=6, 6, 5) | 2068.13 (1008.064) | 2437.78 (949.142) | 2031.41 (997.685)

11. Secondary Outcome: CL/F: Apparent Oral Clearance of MLN3126 and Its Metabolite After Multiple Dosing (at Steady State)
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Day 1: predose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: liter per hour (L/hr)
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
liter per hour (L/hr)
  MLN3126 | 4.76 (0.740) | 7.64 (1.989) | 3.87 (1.132)
  M-I | NA (NA) — As pre-specified in protocol, oral clearance was only calculated for parent drug (MLN3126) and not for metabolite (M-I), hence data is reported for only MLN3126. | NA (NA) — As pre-specified in protocol, oral clearance was only calculated for parent drug (MLN3126) and not for metabolite (M-I), hence data is reported for only MLN3126. | NA (NA) — As pre-specified in protocol, oral clearance was only calculated for parent drug (MLN3126) and not for metabolite (M-I), hence data is reported for only MLN3126.

12. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
hours
  Day 1 (MLN3126) (n=6, 6, 6) | 12.901 (0.9029) | 13.717 (0.9151) | 12.830 (1.9144)
  Day 15 (MLN3126) (n=6, 6, 5) | 13.459 (0.5482) | 12.308 (0.9315) | 12.727 (1.0056)
  Day 1 (M-I) (n=6, 6, 6) | 14.901 (2.7546) | 13.131 (2.9209) | 13.374 (4.6494)
  Day 15 (M-I) (n=6, 6, 5) | 16.644 (3.2368) | 13.724 (2.0905) | 15.086 (3.2709)

13. Secondary Outcome: Cav: Average Plasma Concentration for MLN3126 and Its Metabolite on Day 1
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Day 1: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  MLN3126 | 892.89 (135.079) | 1727.16 (430.824) | 1139.34 (263.254)
  M-I | 84.46 (43.261) | 122.32 (49.186) | 71.74 (32.035)

14. Secondary Outcome: Cavss: Average Plasma Concentration for MLN3126 and Its Metabolite at Steady State on Day 15
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Day 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 5
ng/mL
  MLN3126 | 656.20 (151.354) | 1098.04 (234.426) | 756.95 (188.168)
  M-I | 70.75 (35.716) | 80.00 (28.723) | 68.09 (35.408)

15. Secondary Outcome: Rac AUC(0-96): Accumulation Ratio of AUC(0-96) for MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
ratio
  MLN3126 | 0.66572 (0.084399) | 0.60172 (0.082195) | 0.64024 (0.077509)
  M-I | 0.84423 (0.113307) | 0.65535 (0.100968) | 0.89068 (0.090814)

16. Secondary Outcome: Cmax Ratio: Ratio of Maximum Plasma Concentration Between MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
ratio
  Day 1 | 0.0781 (0.02078) | 0.0732 (0.02842) | 0.0595 (0.01627)
  Day 15 | 0.0774 (0.02228) | 0.0578 (0.01890) | 0.0663 (0.02617)

17. Secondary Outcome: Ratio of AUC(0-tau): Ratio of Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Between MLN3126 and Its Metabolite
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 6 | 6 | 6
ratio
  Day 1 | 0.0909 (0.03620) | 0.0722 (0.02894) | 0.0621 (0.01972)
  Day 15 | 0.1055 (0.04173) | 0.0727 (0.02549) | 0.0898 (0.04073)

18. Secondary Outcome: Ae (0-4): Amount of MLN3126 and Its Metabolite Excreted in Urine From 0 to 4 Hours Post Dose
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 4 hours) post-dose
Population: Data is not reported because the study was terminated early at Cohorts 2A and 1B, yielding limited data for only 2 dose levels of MLN3126 in non-Japanese participants and one dose level in Japanese participants. Therefore the analyses to determine urine PK parameters was not performed.
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Fe (0-4): Fraction of Dose of MLN3126 and Its Metabolite Excreted Unchanged in Urine From 0 to 4 Hours Post Dose
Description: M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 4 hours) post-dose
Population: as for outcome 18
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: CLr: Renal Clearance of MLN3126 and Its Metabolite
Description: CLr is the volume of plasma from which the drug is completely removed by the kidney in a given amount of time, calculated as the amount of drug excreted in the urine divided by the area under the plasma concentration-time curve, expressed in liter per hour (L/hr). M-I is the inactive metabolite of MLN3126.
Time Frame: Days 1 and 15: pre-dose and at multiple timepoints (up to 96 hours) post-dose
Population: as for outcome 18
Arm/Group | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: MLN3126 100 mg
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 7 days after the last dose of double-blind study drug (Day 22 in each part).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part A: Placebo | Part A: MLN3126 100 mg | Part A: MLN3126 300 mg | Part B: Placebo | Part B: MLN3126 100 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/6 | 0/6 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 1/3 | 1/6 | 1/6 | 0/2 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=3) | Part A: MLN3126 100 mg (N=6) | Part A: MLN3126 300 mg (N=6) | Part B: Placebo (N=2) | Part B: MLN3126 100 mg (N=6)
Headache (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be made without Sponsor's prior written approval. Any proposed publication or presentation will be submitted to Sponsor for review 60 days in advance of publication. Institution will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for an additional 60 days to preserve intellectual property.